CLINICAL TRIAL: NCT00005157
Title: Speech Characteristics in Coronary Heart Disease
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1029; R01HL033737 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2000-05

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Coronary Disease
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Coronary Disease

SUMMARY:
To improve the predictive validity of Structured Interview assessments of Type A behavior by comparing interviewer techniques in the Multiple Risk Factor Intervention Trial (MRFIT) and the Western Collaborative Group Study (WCGS). To assess whether there were interviewer differences in the predictiveness of Type A behavior and its components for coronary heart disease incidence in MRFIT and WCGS and if so, to assess whether the interviewer differences in disease predictiveness were related to interviewer stylistics.

DETAILED DESCRIPTION:
BACKGROUND:

Individuals with Type A behavior are characterized as hard driving, competitive, and time urgent; when asked questions they are quick to answer with emphatic speech; they perceive themselves to be striving and competing and are prone to hostility. This core of behaviors is presumed to be on a continuum of intensity with well-developed Type A's at the upper end and well-developed Type B's at the lower end. Epidemiological studies have shown Type A's to have a higher prevalence and incidence of various forms of coronary heart disease than Type B's. The Structured Interview is a method of measuring Type A behavior in which a series of questions are administered about the individual's characteristic responses to situations relevant to the Type A behavior pattern, such as reaction to delay and reported frequency of anger. The Interview is delivered in challenging style designed to elicit Type A characteristics.

In 1960, the WCGS recruited 3,154 employed men, ages 39 to 59, who were initially free of coronary heart disease and followed them for 8.5 years for coronary heart disease incidence. In 1972 MRFIT began recruiting 12,866 men, ages 35 to 57, selected for elevation of one or more risk factors, but free from coronary heart disease and followed them for an average of seven years after randomization to a risk factor modification group or to a control group referred to their own physicians for treatment. Both studies used the Structured Interview to assess Type A behavior.

In 1981, Type A behavior was officially regarded as an independent risk factor for coronary heart disease, based largely on the findings of the WCGS. However, the MRFIT did not find Type A behavior to be related to coronary heart disease incidence. The manner of conducting the Structured Interview may have affected the predictive reliability of the Type A assessments.

DESIGN NARRATIVE:

Interviewer speech characteristics from the WCGS and MRFIT Structured Interview tape recordings were audited and analyzed. Each speech characteristic was scored with high reliability. Multiple logistic regression analyses were used to control for standard risk factors.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1982-07; Study Completion 1989-11 (Actual)

REFERENCES:
- [Background] Scherwitz LW, Evans LA, Hennrikus DJ, Vallbona C. Procedures and discrepancies of blood pressure measurements in two community health centers. Med Care. 1982 Jul;20(7):727-38. doi: 10.1097/00005650-198207000-00008. PMID 7121092
- [Background] Ornish D, Scherwitz LW, Doody RS, Kesten D, McLanahan SM, Brown SE, DePuey E, Sonnemaker R, Haynes C, Lester J, McAllister GK, Hall RJ, Burdine JA, Gotto AM Jr. Effects of stress management training and dietary changes in treating ischemic heart disease. JAMA. 1983 Jan 7;249(1):54-9. PMID 6336794
- [Background] Scherwitz L, McKelvain R, Laman C, Patterson J, Dutton L, Yusim S, Lester J, Kraft I, Rochelle D, Leachman R. Type A behavior, self-involvement, and coronary atherosclerosis. Psychosom Med. 1983 Mar;45(1):47-57. doi: 10.1097/00006842-198303000-00007. PMID 6844528
- [Background] Scherwitz L, Graham L, Ornish D: Self-Involvement and the Risk Factors for Coronary Heart Disease. Advances, Institute for the Advancement of Health. Vol 2:6-18, 1985
- [Background] Scherwitz L, Graham LE 2nd, Grandits G, Buehler J, Billings J. Self-involvement and coronary heart disease incidence in the multiple risk factor intervention trial. Psychosom Med. 1986 Mar-Apr;48(3-4):187-99. doi: 10.1097/00006842-198603000-00004. PMID 3704083
- [Background] Scherwitz L, Graham LE 2nd, Grandits G, Billings J. Speech characteristics and behavior-type assessment in the Multiple Risk Factor Intervention Trial (MRFIT) structured interviews. J Behav Med. 1987 Apr;10(2):173-95. doi: 10.1007/BF00846425. PMID 3612777
- [Background] Scherwitz L, Canick J: Self-Reference and Coronary Heart Disease Risk. In: Houston K & Snyder CR (Eds.), Type A Behavior Pattern: Research, Theory, and Intervention. John Wiley & Sons, New York, 1987
- [Background] Scherwitz L: Interviewer Behaviors in the Western Collaborative Group Study and the Multiple Risk Factor Intervention Trial Structured Interviews. In: Houston K & Snyder CR (Eds.), Type A Behavior Pattern: Research, Theory, and Intervention. John Wiley & Sons, New York, 1987
- [Background] Scherwitz L: Type A Behavior Assessment in the Structured Interview: Review, Critique, and Recommendations. In: Siegman A (Ed.), In Search of Coronary-Prone Behavior. Lawrence Erlbaum, Hillsdale, NJ, 1987
- [Background] Graham LE 2nd, Scherwitz L, Brand R. Self-reference and coronary heart disease incidence in the Western Collaborative Group Study. Psychosom Med. 1989 Mar-Apr;51(2):137-44. doi: 10.1097/00006842-198903000-00003. PMID 2710908
- [Background] Scherwitz L, Graham LE 2nd, Grandits G, Billings J. Speech characteristics and coronary heart disease incidence in the multiple risk factor intervention trial. J Behav Med. 1990 Feb;13(1):75-91. doi: 10.1007/BF00844900. PMID 2348450